CLINICAL TRIAL: NCT02310594
Title: The Effect of Radiation Therapy on Tumor Immunity
Brief Title: Anti-tumor Immune Response in Patients With Cancer Undergoing Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-001588; NCI-2014-02231 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-001588-CR-00004 (Other: Jonsson Comprehensive Cancer Center); Steinberg122308; 09-01-010 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2014-11-13; First posted 2014-12-08 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-01

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The tentative assumption is that cell death following radiation therapy will stimulate anti-tumor immunity, which could provide a more permanent solution to curing cancer and discouraging tumors from spreading throughout the body. In order to find out if this assumption is correct, highly developed, laboratory analyses for tumor-specific immunity will be performed using the white blood cells, while the blood components that are soluble, will be frozen and stored, to be examined at a later time for evidence of molecules of anti-tumor immunity that have been induced by radiation therapy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (blood banking): Samples of blood are collected before, during, and within two weeks after radiation therapy and then stored for analysis of anti-tumor immunity.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: cytology specimen collection procedure — Undergo blood sample collection
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies the effect of radiation therapy on tumor immunity. Standard radiation therapy destroys tumor cells. In response to tumor cell death caused by radiation therapy, the body has an ability to stimulate an anti-tumor response (immunity), but this response is often ineffective in shrinking tumor tissue. Collecting samples of blood from patients before, during, and after radiation therapy to study in the laboratory may help doctors learn more about the effects of radiation therapy on anti-tumor response.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effect of radiation therapy on tumor immunity.

OUTLINE:

Samples of blood are collected before, during, and within two weeks after radiation therapy and then stored for analysis of anti-tumor immunity.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Institutional Review Board (IRB)-approved Informed Consent form for the study
* Received an explanation of the study, including satisfactory answers to all questions related to the proposed research
* Is undergoing physician directed radiation treatment

Exclusion Criteria:

* The potential Subject is unwilling or hesitant to participate for any reason and/or fails to complete the appropriate Informed Consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients undergoing physician directed radiation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2010-07-08 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Outcome measures include changes in tumor-specific immune responses and general immune signature in patients undergoing Radiation Treatment. Reportable endpoints are absolute values of and changes in innate & adaptive immune cells and serum markers. | The time line of interest covers a baseline, pre-treatment sample as well as mid-treatment and a post-treatment, follow-up sample at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Steinberg, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States